CLINICAL TRIAL: NCT01143662
Title: A Multi-center, Randomized, Open-label and Positive Controlled Phase II Clinical Trial to Assess Efficacy and Safety of Ypeginterferon Alfa-2b in HBeAg Positive Patients With Chronic Hepatitis B
Brief Title: Efficacy and Safety of Ypeginterferon Alfa-2b in HBeAg Positive Chronic Hepatitis B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TB1007IFN
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Hepatitis B
Keywords: peginterferon; interferon; Pegasys; HBV; Hepatitis B; HBeAg positive
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): Ypeginterferon alfa-2b 90mcg per week
  Interventions: Drug: Ypeginterferon alfa-2b
- Group 2 (Experimental): Ypeginterferon alfa-2b 135mcg per week
  Interventions: Drug: Ypeginterferon alfa-2b
- Group 3 (Experimental): Ypeginterferon alfa-2b 180mcg per week
  Interventions: Drug: Ypeginterferon alfa-2b
- Group 4 (Active Comparator): Pegasys 180mcg per week
  Interventions: Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Ypeginterferon alfa-2b — sc, qw, for 48 weeks.
  Arms: Group 1; Group 2; Group 3
Drug: Peginterferon alfa-2a — sc, qw, for 48 weeks.
  Other Names: Pegasys
  Arms: Group 4

SUMMARY:
This study is a multi-center, randomized, open-label and positive controlled Phase II Clinical trial to assess efficacy and safety of Ypeginterferon alfa-2b, once a week, in 3 dose-groups: 90mcg, 135mcg and 180mcg, respectively, for treatment of chronic hepatitis B characterized by HBeAg positivity, with Pegasys 180mcg/week as positive control. It is aimed to establish a dose response and safety relationship sufficient to allow the subsequent design and conduct of Phase III trials, and generate pharmacokinetic data of Ypeginterferon alfa-2b in hepatitis B patients to satisfy regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Age:18~60 years.
* Pregnancy tests of female patients must be negative. All patients with effective birth control measures during treatment period and 6 months after the cessation of treatment.
* Serum HBsAg positive for at least 6 months.
* Serum HBeAg positive with HBV DNA ≥20,000IU/ml.
* 2×ULN≤ALT≤10×ULN at screening(ULN=upper limit of normal).

Exclusion Criteria:

* Pregnant or lactating women.
* Mental disorder or physical disability.
* Interferon treatment history or using nucleos(t)ide analogue for chronic hepatitis B treatment within the previous 6 months.
* WBC<3000/mm3, or ANC <1500/mm3, or PLT <90,000/mm3.
* Co-infection with HAV, HIV, HCV, HDV, HEV.
* Both HBsAg and anti-HBs are positive, or both HBeAg and anti-HBe are positive at screening.
* Chest X-ray with clinically significant active inflammatory process, history of significant pulmonary disease or any history of interstitial lung disease.
* Evidence of hepatic decompensation.
* History of hypothyroidism or current treatment for thyroid disease.
* Uncontrolled significant chronic medical conditions other than chronic hepatitis B, or other conditions which in the opinion of the investigator preclude enrollment into the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 205 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Efficacy | week 24 from treatment start
  * Average of HBV DAN decline level at week 24.
  * Proportion of patients with HBeAg undetectable and HBeAg seroconversion at week 24.

SECONDARY OUTCOMES:
Efficacy | week 12, 24, 48 from treatment start and week 24 after treatment
  * Average of HBV DNA decline level at week 12, 48 and 72.
  * Proportion of patients with HBV DNA undetectable at week 48 and 72.
  * Proportion of patients with HBeAg undetectable and HBeAg seroconversion at week 48 and 72.
  * Proportion of patients with HBsAg undetectable and HBsAg seroconversion at week 48 and 72.
  * Proportion of patients with ALT normalization at week 24 and 48.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Guiqiang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (39):
- China (39):
  - 302 Military Hospital, Beijing
  - Beijing Youan Hospital, Capital Medical University, Beijing
  - Beijing Youyi Hospital, Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - First Affiliated Hospital of Jilin University, Changchun
  - Xiangya Hospital, Central-south University, Changsha
  - Xiangya Second Hospital, Central-south University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - Southwest Hospital, Chongqing
  - Fuzhou Infectious Disease Hospital, Fuzhou
  - Guangzhou Eighth People's Hospital, Guangzhou
  - Nanfang Hospital, Guangzhou
  - Third Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - First Affiliated Hospital of Guangxi Medical University, Guilin
  - First Affiliated Hospital, Zhejiang University, Hangzhou
  - Second Affiliated Hospital of Harbin Medical University, Harbin
  - First Affiliated Hospital of Anhui Medical University, Hefei
  - Jinan Infectious Disease Hospital, Jinan
  - First Affiliated Hospital of Lanzhou University, Lanzhou
  - First Affiliated Hospital of Nanchang University, Nanchang
  - 81 Military Hospital, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - Second Hospital of Nanjing, Nanjing
  - 85 Militay Hospital, Shanghai
  - Changhai Hospital, Shanghai
  - Huashan Hospital, Shanghai
  - Renji Hospital, Shanghai
  - Ruijin Hospital, Shanghai
  - Shanghai Public Health Clinical Center, Shanghai
  - Shenzhen Third People's Hospital, Shenzhen
  - Third Affiliated Hospital, Hebei Medical University, Shijiazhuang
  - First Affiliated Hospital, Shanxi University, Taiyuan
  - Tianjin Third Central Hospital, Tianjin
  - First Affiliated Hospital of Wenzhou Medical College, Wenzhou
  - Tongji Hospital, Huazhong University of Science&Technology, Wuhan
  - Tangdu Hospital, Fourth Military Medical University, Xi'an
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Henan Provincial People's Hospital, Zhengzhou